CLINICAL TRIAL: NCT04756817
Title: Immunogenicity of the BNT162b2 mRNA Covid-19 Vaccine in Elderly People Over 85 Years of Age: Real World Data From Greece
Brief Title: Immunogenicity of the BNT162b2 Covid-19 Vaccine in Elderly People Aged 85 and Older in Greece
Acronym: GREVAXIMO
Status: Completed | Type: Observational
Sponsor: G.Gennimatas General Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgios Papazisis, Associate Professor of Clinical Pharmacology, Aristotle University Of Thessaloniki
Other Study IDs: 2/27.1.2021
Record Dates: First submitted 2021-02-14; First posted 2021-02-16 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Immunogenicity, Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples retained, with no potential for DNA extraction from any retained sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Real-world evidence confirming the effectiveness and safety of the new COVID-19 vaccines among the elderly is currently lacking. However, scarce (sparse) data derived from phase II/III trials attest to a weaker humoral immune response generated post-immunization among seniors, in contrast to younger adults. According to the national priority vaccination scheme the age group of 85 and older was the first to receive the BNT162b2 mRNA Covid-19 vaccine in Greece. The aim of the study is to enhance our insight into the humoral immunity and antibody generation elicited by the BNT162b2 mRNA Covid-19 vaccine among the elderly. The study population will include people aged 85 or older who are either uninfected or have a positive history of PCR-confirmed SARS-CoV-2 infection occurring one to 4.5 months prior to vaccination. Upon receipt of informed consent, a cohort of persons vaccinated in the two vaccination centers of the "G. Gennimatas" General Hospital of Thessaloniki will be followed over a period of six months post-injection of the second dose. To monitor the immunogenicity of the BNT162b2 mRNA Covid-19 vaccine, the SARS-CoV-2 IgG II Quant assay will be applied to conduct both qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein on day 21 after the first dose, day 21 after the second dose and within 3 and 6 months after the second dose.

DETAILED DESCRIPTION:
Real world data regarding the effectiveness and safety of the new COVID-19 vaccines in older people are currently lacking. The sparse data from Phase II/II trials suggest a reduction in antibody responses in older people compared to younger participants. The over-85 age group was the first group to receive the BNT162b2 mRNA Covid-19 vaccine in Greece according to the national priority vaccination scheme. The aim of the study is to enhance insight into the immunity and antibody generation elicited by the BNT162b2 mRNA Covid-19 vaccine among elderly people over age 85. The study population will include both uninfected vaccinated persons and persons with PCR-confirmed previous SARS-CoV-2 infection occurring one to 4.5 months prior to vaccination. After informed consent a cohort of persons vaccinated in the two vaccination centers of the "G. Gennimatas" General Hospital of Thessaloniki will be followed for six months post-second dose injection. The immunogenicity of the vaccine will be measured using the SARS-CoV-2 IgG II Quant assay to conduct a qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein on day 21 after the first dose, day 21 after the second dose and within 3 and 6 months after the second dose.

Having set the positivity threshold of the immunoassay (50 AU/ml) as a cut-off point, participants will be classified both by history of infection with SARS-CoV-2 and by SARSCoV-2 IgG II Quant assay outcomes. Subsequently, the IgG geometric mean concentration (GMC) and its 95% Confidence Interval will be calculated, based on the recorded antibody concentration values. Regarding the reactogenicity of the vaccine, on the day of blood collection the participants will be asked to report their experienced side effects. Of note, participants are asked to officially report all unsolicited adverse drug reactions (ADRs) to the National Medicines Organization via the Yellow Card scheme. The study protocol has been endorsed and ethical approval was obtained by the ethics committee of the scientific council of the "G. Gennimatas" General Hospital (protocol number:2/12.02.2021).

Regarding the reactogenicity of the vaccine, on the day of blood collection the participants will be asked to report their experienced side effects. Of note, participants are asked to officially report all unsolicited adverse drug reactions (ADRs) to the National Medicines Organization via the Yellow Card scheme.

The study protocol was approved and ethical approval was obtained by the ethics committee of the scientific council of the "G. Gennimatas" General Hospital (protocol number:2/12.02.2021).

ELIGIBILITY:
Inclusion Criteria:

1. Age of 85 or older
2. Without previously known SARS-CoV-2 infection, or
3. With previous PCR-confirmed SARS-CoV-2 infection one to 4.5 months prior to vaccination

Exclusion Criteria:

* Occurence of any other vaccination 4 weeks prior to enrollment
* Participation in any other clinical trial

Ages: 85 Years to 100 Years | Sex: All
Age Groups: Older Adult
Study Population: Elderly aged 85 or older prioritised for vaccination based on the greek national vaccination plan
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2021-02-13 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Immunogenicity after the first dose of the BNT162b2 mRNA Covid-19 vaccine | 21 days after the first dose
  Immunogenicity of the BNT162b2 mRNA Covid-19 vaccine measured using the SARS-CoV-2 IgG II Quant assay to conduct a qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein on day 21 after the first dose
Immunogenicity after the second dose of the BNT162b2 mRNA Covid-19 vaccine | 21 days after the second dose
  Immunogenicity of the BNT162b2 mRNA Covid-19 vaccine measured using the SARS-CoV-2 IgG II Quant assay to conduct a qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein on day 21 after the second dose
Immunogenicity after the second dose of the BNT162b2 mRNA Covid-19 | 3 months after the second dose
  Immunogenicity of the BNT162b2 mRNA Covid-19 vaccine measured using the SARS-CoV-2 IgG II Quant assay to conduct a qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein 3 months after the second dose
Immunogenicity after the second dose of the BNT162b2 mRNA Covid-19 | 6 months after the second dose
  Immunogenicity of the BNT162b2 mRNA Covid-19 vaccine measured using the SARS-CoV-2 IgG II Quant assay to conduct a qualitative and quantitative determination of IgGs against the receptor-binding domain (RBD) of the S1 subunit of the SARS-CoV-2 spike protein 6 months after the second dose

SECONDARY OUTCOMES:
PCR-confirmed cases of SARS-CoV-2 infection anytime after the first dose. | 6 months after the second dose
  PCR-confirmed cases of SARS-CoV-2 infection anytime after the first dose measured using hospital records

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Papazisis, As.Professor, Study Chair — School of Medicine,Aristotle University of Thessaloniki
Locations (1):
- G. Gennimatas General Hospital, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study will be available from the corresponding author on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and any additional supporting information will become available starting 6 months after publication
Access Criteria: Completely anonymised, de-identified (stripped of all "direct identifiers") numerical data in spreadsheets will be shared with researchers from the academia and relevant research institutions after the publication of corresponding results in peer reviewed academic journals, for purposes of independent statistical analysis and verification of results. Participants will provide consent for the use of anonymised data for research purposes.

REFERENCES:
- [Background] Kontopoulou K, Nakas CT, Ainatzoglou A, Ifantidou A, Ntotsi P, Katsioulis C, Papazisis G. Immunogenicity of the BNT162b2 mRNA Covid-19 vaccine in elderly people over 85 years of age in Greece: the GREVAXIMO study. Aging Clin Exp Res. 2021 Dec;33(12):3385-3389. doi: 10.1007/s40520-021-01997-7. Epub 2021 Oct 11. PMID 34633648